CLINICAL TRIAL: NCT05382533
Title: Modulation of Cardiovascular Risk II (MoKaRi II) Intervention Study - Modulation of Cardiovascular Risk and Diabetes Risk Using Menu Plans
Brief Title: MoKaRi II Intervention Study
Acronym: MoKaRi II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Christine Dawczynski,PhD, PhD, University of Jena
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H13-22
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Decreased Cardovascular Risk; Decreased Risk of Diabetes Mellitus Type II
Keywords: triacylglcerides, glucose, HbA1c, body weight
MeSH Terms: conditions — Body Weight | interventions — Menu Planning

STUDY DESIGN:
Intervention Model Description: parallel design
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hypertriglyceridemia intervention (group A) (Experimental): * Carbohydrates: ≤ 50 en% (sucrose + glucose + fructose ≤ 10 en%, where sucrose ≤ 5 en% and fructose ≤ 20 g/d)
  * Fat: 30-35 En%
  * Protein: 20 En%
  * marine n3 PUFA (EPA/DHA): ≥ 4000 mg/d (10 g fish oil)
  Interventions: Dietary Supplement: Menu plans
- Hypertriglyceridemia control (group B) (No Intervention): no menu plans, no study foods
- Prediabetes intervention (group C) (Experimental): * Carbohydrates: 40 ± 2 En%
  * Sucrose + glucose + fructose ≤ 10 En%
  * Free sugars < 5% of daily energy
  * Fat: 40 ± 2%
  * Protein: 20 ± 2 En%
  * n3 PUFA: ≥ 500 mg/d
  Interventions: Dietary Supplement: Menu plans
- Prediabetes control (group D) (No Intervention): no menu plans, no study foods

INTERVENTIONS:
Dietary Supplement: Menu plans — The study participants in group A and C receive defined personal nutritional counselling every two weeks and they are provided with daily menu plans (isocaloric) with optimized nutrient profiles and chosen study products (plant oils, nuts mixture etc.) over the study period of 10 weeks.
  Arms: Hypertriglyceridemia intervention (group A); Prediabetes intervention (group C)

SUMMARY:
The proposed intervention study addresses the development and validation of nutritional concepts based on menu plans for patients with hypertriglyceridemia (triglycerides > 1.5 mmol/l) and participants with impaired glucose tolerance/prediabetes (glucose > 5.6 ≤ 7 mmol/l).

DETAILED DESCRIPTION:
The proposed intervention study addresses the development and validation of nutritional concepts for patients with hypertriglyceridemia (triglycerides > 1.5 mmol/l) and participants with impaired glucose tolerance (glucose > 5.6 ≤ 7 mmol/l).

The randomized, controlled study will be conducted in a parallel design with four arms. In total, 120 participants (males, females; age: 30 - 80 years) will be randomized to one of the four groups: hypertriglyceridemia concept (group A), hypertriglyceridemia control (group B), prediabetes concept (group C), and prediabetes control (group D).

The study participants in group A and C receive defined personal nutritional counselling every two weeks and they are provided with daily menu plans (isocaloric) with optimized nutrient profiles and chosen study products (e.g., fish or plant oil, nuts) over the study period of ten weeks. Participants in the control groups B and D are not provided with defined menu plans or study products.

Blood samples will be taken at the beginning, regularly every two weeks of the ten-weeks intervention period as well as after the ten-weeks follow-up. Primary endpoints are triglycerides (group A, B), and fasting glucose (group C, D).

The study design enables the comparison of the effectiveness of the developed nutritional concepts, which were adapted to the requirements of the target groups.

ELIGIBILITY:
Inclusion Criteria:

Voluntary participation with documented consent

* Willingness and ability to adhere to study protocol
* Volunteer test person (m/f) aged ≥ 30 years and ≤ 80 years
* BMI: ≥ 20 ≤ 40 kg/m2
* No or moderate alcohol consumption (≤ 2 glasses/week)
* non-smoker (if possible)
* Group A, B: triglycerides: > 1.5 mmol/l
* Group C, D: Fasting glucose: ≥ 5.6 ≤ 7 mmol/L

Exclusion Criteria:

Concomitant diseases:

* Hypercholesterolemia (genetic defect / familial predisposition)
* Diabetes mellitus
* Thyroid dysfunction (hyper- or hypothyroidism)
* Food intolerances/allergies to ingredients in the study foods
* Medications: lipid-lowering drugs, glucocorticoids, oral medication for the treatment of type 1-4 diabetes mellitus, insulin injections
* Dietary supplements: especially n-3 fatty acids, vitamin E
* Extremely high physical activity (daily)
* Alcohol abuse (daily)
* (smokers) [if there are not enough subjects available, at least 7 smokers should be included so that a statistical analysis is possible]
* Uncontrolled organic diseases
* Alcohol, medication or drug abuse
* Participation in other observational clinical studies during or 4 wk. before starting this study
* Severe behavioral, emotional, or psychiatric problems that the investigator determined would result in non-compliance
* Pregnancy, lactation and unsafe contraception
* Other reasons considered important by the investigator

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Triacylglcerides, mmol/l (group A, B) | Change from baseline after 10 weeks
  Cardiovascular risk factor
Fasting glucose, mmol/l (group C, D) | Change from baseline after 10 weeks
  Diabetes risk factor

SECONDARY OUTCOMES:
Total cholesterol (mmol/l) | Change from baseline after 10 weeks
  Cardiovascular risk factor
HDL cholesterol (mmol/l) | Change from baseline after 10 weeks
  Cardiovascular risk factor
LDL cholesterol (mmol/l) | Change from baseline after 10 weeks
  Cardiovascular risk factor
Systolic pressure (mm Hg) | Change from baseline after 10 weeks
  Cardiovascular risk factor
Diastolic pressure (mm Hg) | Change from baseline after 10 weeks
  Cardiovascular risk factor
Insulin (mU/l) | Change from baseline after 10 weeks
  Diabetes risk factor
HbA1c (%) | Change from baseline after 10 weeks
  Diabetes risk factor
Body weight (kg) | Change from baseline after 10 weeks
  Cardiovascular risk factor
Body fat (kg) | Change from baseline after 10 weeks
  Cardiovascular risk factor
High sensitive c-reactive protein (mg/l) | Change from baseline after 10 weeks
  Inflammatory marker
Fatty acid distribution in erythrocyte lipids (% fatty acid methyl esters) | Change from baseline after 10 weeks
  Fatty acid distribution in erythrocyte lipids
Vitamin A (mmol/l) | Change from baseline after 10 weeks
  Vitamins
Vitamin D (nmol/l) | Change from baseline after 10 weeks
  Vitamins
Vitamin E (µmol/l) | Change from baseline after 10 weeks
  Vitamins
Vitamin B1 (nmol/l) | Change from baseline after 10 weeks
  Vitamins
Vitamin B6 (nmol/l) | Change from baseline after 10 weeks
  Vitamins
Vitamin B12 (pmol/l) | Change from baseline after 10 weeks
  Vitamins
Holo-transcobalamin (pmol/l) | Change from baseline after 10 weeks
  Vitamins
Folic acid (µg/l) | Change from baseline after 10 weeks
  Vitamins
Vitamin H (ng/l) | Change from baseline after 10 weeks
  Vitamins
Vitamin C (mg/l) | Change from baseline after 10 weeks
  Vitamins
Potassium (mmol/l) | Change from baseline after 10 weeks
  Minerals and trace elements
Iron (µmol/l) | Change from baseline after 10 weeks
  Minerals and trace elements
Ferritin (µg/l) | Change from baseline after 10 weeks
  Minerals and trace elements
Transferrin (g/l) | Change from baseline after 10 weeks
  Minerals and trace elements
Iodine (µmol/l) | Change from baseline after 10 weeks
  Minerals and trace elements
Selenium (µmol/l) | Change from baseline after 10 weeks
  Minerals and trace elements
Zinc (µmol/l) | Change from baseline after 10 weeks
  Minerals and trace elements

OTHER OUTCOMES:
Creatinine (mmol/l) | Change from baseline after 10 weeks
  Creatinine (24 h urine)
Albumine (mg/l) | Change from baseline after 10 weeks
  Albumine (24 h urine)
Selenium (µmol/24 h) | Change from baseline after 10 weeks
  Selenmium (24 h urine)
Zinc (µmol/24 h) | Change from baseline after 10 weeks
  Zinc (24 h urine)

CONTACTS AND LOCATIONS:
Overall Officials: Christine A Dawczynski, PhD, Principal Investigator — Friedrich Schiller University Jena
Locations (1):
- Institute of Nutritional Sciences, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.nuco.uni-jena.de/studien